CLINICAL TRIAL: NCT05640817
Title: Clinical Study Evaluating the Nephroprotective Effect of Pentoxifylline Against Cisplatin in Patients With Head and Neck Cancer
Brief Title: Nephroprotective Effect of Pentoxifylline Against Cisplatin in Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eman Elberri, Lecturer of Clinical Pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PTX122022
Record Dates: First submitted 2022-11-30; First posted 2022-12-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pentoxifylline, Cisplatin, Nephrotoxixcity
MeSH Terms: interventions — Pentoxifylline; Cisplatin; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 as control group (Active Comparator): cisplatin with standard hydration with normal saline
  Interventions: Drug: cisplatin with standard hydration with normal saline
- Group two as Pentoxifylline (Active Comparator): receive cisplatin with standard hydration with normal saline and Pentoxifylline 400 mg SR tablets twice daily for three cycles.
  Interventions: Drug: Pentoxifylline 400 mg SR tablets

INTERVENTIONS:
Drug: Pentoxifylline 400 mg SR tablets — a nonspecific phosphodiesterase inhibitor, was first considered in the treatment of peripheral vascular diseases
  Arms: Group two as Pentoxifylline
Drug: cisplatin with standard hydration with normal saline — chemotherapy
  Arms: Group 1 as control group

SUMMARY:
Head and neck squamous cell carcinoma (HNSCC) encompasses a variety of tumors originating in the lip, oral cavity, hypopharynx, oropharynx, nasopharynx and larynx. It is the sixth most common malignancy worldwide accounting for approximately 6% of all cancer cases (Rettig and D'Souza., 2015). HNSCC represents the third most common cause of cancer death worldwide. Platinum based regimens represent cornerstone in its treatment (Galbiattiet al., 2013).

Cisplatin (cis-diammine dichloroplatinum (II), CDDP) is an inorganic platinum-based chemotherapeutic agent that is widely used in treatment of various solid malignancies as head and neck, lung, testis, ovarian, and bladder cancers (Aparecida et al., 2012). The use of cisplatin is frequently limited by significant side effects including bone marrow suppression, peripheral neuropathy, ototoxicity, anaphylaxis and nephrotoxicity with the latter representing the main dose limiting one (Aparecida et al., 2012).

Acute kidney injury (AKI), distal renal tubular acidosis, renal concentrating defect, transient proteinuria, hyperuricemia, Fanconi-like syndrome, hypomagnesemia, hypocalcemia, renal salt wasting, erythropoietin deficiency, thrombotic microangiopathy, and chronic renal failure are among the renal side effects of cisplatin (Miller et al., 2010).Renal function deterioration is seen in 25% to 35% of patients treated with a single dose of cisplatin (Miller et al., 2010).Cisplatin-induced injury to renal epithelial cells results in the production of various inflammatory factors, including TNF-α. Cisplatin also increases ROS production, which leads to the activation of apoptosis and necrosis pathways (Miller et al., 2010).

Pentoxifylline (PTX), a nonspecific phosphodiesterase inhibitor, was first considered in the treatment of peripheral vascular diseases (Nasiri-Toosi et al., 2013). PTX has anti-inflammatory effects as it down regulates several pro-inflammatory cytokines, including tumor necrosis factor alpha (TNF-α) and interleukin-1 (IL-1) and IL-6 (Mostafa-Hedeab et al., 2022). In addition, PTX has gained considerable interest as a reactive oxygen species (ROS) scavenger, and several studies show its potential antioxidant effects (Zhang et al., 2016). Several studies evaluate the renoprotective effects of PTX against drug-induced nephrotoxicity (Ramesh and Reeves, 2002; Kasap et al., 2013;Nasiri-Toosi et al.,2013; Panahi-Shokouh etal., 2020; Alorabi et al., 2022).

ELIGIBILITY:
Inclusion criteria:

1. Patient aged 18 years or more with head and neck cancer who will receive cisplatin for the first time.
2. Baseline estimated glomerular filtration rate (eGFR) ≥ 59 ml/min/1.73 m2.
3. Eastern Cooperative Oncology Group performance status (ECOG) < 2.
4. Patients with normal organic function as defined for the following criteria:

   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 times the upper normal limit of the local laboratory ;
   * Total serum bilirubin ≤ 2.0 x ULN-LL;
   * Absolute neutrophil count ≥ 1,500 / mm3;
   * Platelet count ≥ 100,000 / mm3;
   * Hemoglobin ≥ 8.0 g / dl;
   * Serum creatinine ≤ 1.5 x ULN-LL

Exclusion criteria:

1. Pregnant or nursing women, or females intending pregnancy were all prohibited
2. Patients with concurrent other malignancy or history of other malignancy treated within the past 3 years.
3. Baseline estimated glomerular filtration rate (eGFR) < 59 ml/min/1.73 m2.
4. Alanine aminotransferase (ALT) > 3× times ULN.
5. Eastern Cooperative Oncology Group performance status (ECOG) ≥2.
6. Patients have Diabetes mellitus.
7. Patients have current participation in other protocols with experimental drugs.
8. Patients with no ability to ingest food orally.
9. Pentoxifylline hypersensitivity.
10. Use of other nephrotoxic drugs as aminoglycosides, non-steroidal anti-inflammatory drugs and contrast media.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
nephrotoxicity improvement as measured by CTACE version 5.0 | up to 6 months

SECONDARY OUTCOMES:
Kidney injury molecule 1 decrease serum level | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt